CLINICAL TRIAL: NCT03967288
Title: The Maternal CLIMB Trial: Chloroprocaine to Reduce the Impact of Motor Block on Patient Recovery After Short Obstetric Surgery
Brief Title: Comparison of Clorotekal and Bupivacaine for Short Obstetric Surgery
Acronym: CLIMB
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Four patients required conversion to GETA (2 in each study arm)
Sponsor: Oregon Health and Science University (Other)
Collaborators: B. Braun Medical Inc. (Industry)
Responsible Party: Principal Investigator, Brandon M Togioka, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB#19846
Record Dates: First submitted 2019-05-26; First posted 2019-05-30 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Anesthesia, Spinal
Keywords: Chloroprocaine; Bupivacaine; Motor Block; Anesthesia, Obstetrical
MeSH Terms: interventions — chloroprocaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The subject, obstetrical provider, investigator, and outcomes assessor will be blinded. The anesthesia provider will be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chloroprocaine (Experimental): 50 mg of 1% spinal chloroprocaine (5 mL) injected into the intrathecal space over approximately 5 seconds once prior to the start of surgery
  Interventions: Drug: Chloroprocaine Injection [Clorotekal]
- Bupivacaine (Active Comparator): 10.5 mg of spinal hyperbaric bupivacaine (1.4 mL of 0.75% bupivacaine hydrochloride in 8.25% dextrose) injected into the intrathecal space over approximately 5 seconds once prior to the start of surgery
  Interventions: Drug: Bupivacaine Hydrochloride 0.75% Injection Solution

INTERVENTIONS:
Drug: Chloroprocaine Injection [Clorotekal] — 1% chloroprocaine Hydrochloride Injection (50 mg/5 mL) for intrathecal use
  Other Names: Clorotekal
  Arms: Chloroprocaine
Drug: Bupivacaine Hydrochloride 0.75% Injection Solution — 0.75% bupivacaine Hydrochloride injection in 8.25% dextrose for intrathecal use
  Other Names: Marcaine spinal
  Arms: Bupivacaine

SUMMARY:
The following obstetric procedures are commonly performed with spinal anesthesia on labor and delivery: bilateral tubal ligation, external cephalic version, cerclage insertion, cerclage removal, minimally invasive fetal surgery, and evacuation of retained products of conception. Bupivacaine is currently the standard spinal medication for these procedures because of its long history of safe use, its low incidence of transient neurologic symptoms, and its ability to provide a dependable, dense block with a high degree of maternal satisfaction. While bupivacaine has the aforementioned advantages, it unfortunately has a long duration of action, up to 240-380 minutes, which far exceeds the time necessary to complete most obstetric procedures. Clorotekal®, the first Food and Drug Administration approved chloroprocaine solution created for spinal injection, is a potential alternative. When compared with bupivacaine spinals, chloroprocaine spinals have been shown to facilitate clinically significant shorter times to resolution of motor and sensory block, first ambulation, micturition, and discharge readiness. The objective of this study is to determine if a strategy of spinal anesthesia with chloroprocaine will reduce the duration of motor block, compared with equivalent block with hyperbaric bupivacaine..

DETAILED DESCRIPTION:
This will be a single-blind, randomized, controlled, single center clinical trial assessing the efficacy of spinal chloroprocaine on resolution of motor block and associated patient flow through the post-anesthesia care unit . Fifty patients will be equally randomized to receive either spinal chloroprocaine or hyperbaric bupivacaine.

Masking:

1. Subject
2. Obstetric provider
3. Investigator
4. Outcomes assessor

The anesthesia provider will be unblinded.

Subjects will be allocated to either intrathecal injection of 50 mg of 1% chloroprocaine or 10.5 mg (1.4 mL) of 0.75% hyperbaric bupivacaine. The intrathecal space will be accessed with a 25 gauge Whitacre needle. Upon obtaining cerebrospinal fluid, the syringe of study solution will be attached the end of the Whitacre needle. The syringe will be pulled back to reveal aspiration of cerebrospinal fluid. The study solution will then be administered over approximately 5 seconds. The Whitacre needle and spinal introducer needle will be removed from the patient's back. The patient will be placed supine on the operating room table. The outcomes assessor will then be allowed to enter the operating room.

Decisions on when to administer additional sedative and analgesic medications will be left to the discretion of the anesthesia team. The level of block will be initially assessed by the anesthesia team. When the block is felt to be at peak height the outcomes assessor will test with pinprick to determine the peak block height.

In accordance with standard of practice at our institution all patients will have convective warmers used during the case and patient temperature will be monitored. Non-invasive blood pressures will be obtained every 2.5 minutes after spinal placement. The frequency of blood pressure measurement will be changed to every 5 minutes, 15 minutes after spinal placement. Anesthesia providers will administer phenylephrine via intravenous bolus to maintain maternal blood pressure within 20% of baseline or for a systolic blood pressure < 100 mm Hg. Anesthesia providers will be allowed to add ephedrine or glycopyrrolate to phenylephrine for maternal hypotension with co-existent bradycardia.

A research coordinator will remain with the patient throughout their time in the operating room and the post-anesthesia care unit. Active, non-standard of care, monitoring for the following signs and symptoms of local anesthetic toxicity will occur in the operating room and post-anesthesia care unit at the following time intervals after spinal placement: 5 minutes, 10 minutes, 15 minutes, upon post-anesthesia care unit arrival, upon completing Phase 1 of post-anesthesia care unit recovery, and upon discharge from the post-anesthesia care unit:

* Seizures
* Tinnitus
* Metallic taste
* Agitation
* Sedation
* Respiratory depression (respiratory rate < 10 breaths per minute)
* Dizziness
* Nausea
* Vomiting
* Vision changes
* Paresthesia
* Perioral numbness
* Hypotension (drop in mean arterial pressure > 20% or systolic blood pressure < 100 mm Hg)
* Arrhythmias

The research coordinator will obtain from anesthesia, upon arrival to the post-anesthesia care unit, the total dose of intraoperative opioids administered, whether the patient had intraoperative hypotension, and the total dose of intraoperative phenylephrine administered. In the post-anesthesia care unit, the research coordinator will determine the patient's Bromage scale score at 5-minute increments. The research coordinator will also ask the patient to notify them when they have a Bromage scale score of 2 (able to flex knees). While in the post-anesthesia care unit, the research coordinator will also document the time of post-anesthesia care unit arrival, the end of Phase 1 of post-anesthesia care unit recovery, and the time that the patient leaves the post-anesthesia care unit (end of Phase 2).

The research coordinator will meet with the patient on the evening of their surgery as well as daily for the duration of their hospitalization to assess for time of first ambulation, bladder catheterization, and for adverse events including, new postoperative neurologic deficits and any other potential adverse events.

To gather information on the incidence of new postoperative neurologic deficits all patients will be called 1 week after spinal insertion. A telephone script will be used to obtain this information.

ELIGIBILITY:
Inclusion Criteria:

1. Women 18 years old to 60 years old
2. American Society of Anesthesiologists physical status class 1-3
3. Undergoing one of the following obstetric procedures: bilateral tubal ligation, external cephalic version, cerclage insertion, cerclage removal, minimally invasive fetal surgery, or evacuation of retained products of conception.

Exclusion Criteria:

1. Refusal of consent
2. Multiple gestations
3. History of ester local anesthetic or para-aminobenzoic acid allergy
4. Height less than 5 feet or greater than 6 feet
5. Body mass index less than 18.5 kg/m2 or greater than 45 kg/m2
6. Any coagulopathy defined by platelets < 80k/microliter, International Normalized Ratio > 1.2, or Partial Thromboplastin Time > 36 seconds
7. Signs of hypovolemia that is not corrected by routine management including hypotension (systolic blood pressure < 90 mm Hg) at the time of evaluation
8. Liver disease including jaundice and ascites, with elevated liver function tests, Aspartate Aminotransferase > 2x institutional normal, Alanine Aminotransferase > 2x institutional normal
9. Renal disease including history of dialysis, with elevated renal function tests on admission labs, glomerular filtration rate < 60 ml/min/1.73 m2
10. Infection at the site of potential spinal insertion
11. Neurologic condition that contraindicates spinal anesthesia, tethered spinal cord or multiple sclerosis
12. Known atypical plasma cholinesterase activity
13. Other contraindications to receive a spinal anesthetic
14. Vulnerable populations including prisoners and decisionally impaired adults

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Motor block-interval assessment | 5 hours
  Bromage scale score at 5 minute intervals, since spinal injection. Interval assessment motor block will be defined as the number of 5-minute intervals since completion of spinal injection to achieve a Bromage score or 2 (able to flex knees)

SECONDARY OUTCOMES:
Motor block-patient report | 5 hours
  The patient will be instructed to notify the outcomes assessor when they are able to flex their knees (Bromage score 2). Patient report motor block will be defined as the time interval in minutes since completion of spinal injection to achieve a Bromage score of 2 (able to flex knees).
Phase 1 Post-Anesthesia Care Unit time | 8 hours
  Phase 1 Post-Anesthesia Care Unit time will be defined as the interval between "out of operating room" and "end of Phase 1" as documented by the Post-Anesthesia Care Unit nurse.
Post-Anesthesia Care Unit time (Phase 1 + Phase 2) | 12 hours
  Post-Anesthesia Care Unit time will be defined as the interval between "out of operating room" and "end of Phase 2" as documented by the labor and delivery nurse for patients discharged home and as mutually agreed upon by the outcomes assessor and nurse for patients discharged to the ward. In addition to meeting Phase 1 criteria, patients must be able to ambulate, micturate, and tolerate food intake in order to exit Phase 2 of Post-Anesthesia Care Unit recovery. Completing Phase 2 of Post-Anesthesia Care Unit recovery is also requires that a responsible adult can escort the patient out of the hospital and remain with the patient for the first 24 hours.
Time to ambulation | 24 hours
  Defined as the time interval in minutes between intrathecal medication administration and time to first ambulation. Ambulation requires a Bromage score of 1 and a standard nursing assessment that is already in practice at Oregon Health and Science University (OHSU).
Bladder Catheterization | 24 hours
  Defined as inserting either a Foley or Straight catheter into the bladder

OTHER OUTCOMES:
Opioid consumption | 2 hours
  Defined as the total intraoperative opioid consumption in milligram morphine equivalents.
Peak block sensory level | 1 hour
  Defined as the most caudal dermatome with sensation to pinprick at the time of "anesthesia ready."

CONTACTS AND LOCATIONS:
Overall Officials: Brandon M Togioka, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU Labor and Delivery; Oregon Health and Science University Hospital, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-19): https://cdn.clinicaltrials.gov/large-docs/88/NCT03967288/Prot_SAP_000.pdf